CLINICAL TRIAL: NCT02285374
Title: A Phase IV Open-label, Multi-centre, Randomised, Dual-arm, Pilot Study to Assess the Feasibility of Switching Individuals Receiving Efavirenz With Continuing Central Nervous System (CNS) Toxicity, to Dolutegravir
Brief Title: Efavirenz to Dolutegravir Switch in Patients With CNS Toxicity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St Stephens Aids Trust (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSAT 056
Record Dates: First submitted 2014-10-13; First posted 2014-11-07 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-10

CONDITIONS: HIV
MeSH Terms: interventions — dolutegravir; efavirenz; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Truvada (tenofovir 245mg/emtricitabine 200mg) or Kivexa (abacavir 600mg/lamivudine 300mg) one tablet once daily plus Dolutegravir 50mg (one tablet) once daily
  Interventions: Drug: Dolutegravir, efavirenz, efavirenz/emtricitabine/tenofovir
- Arm 2 (Experimental): Atripla (efavirenz 600mg, emtricitabine 200mg, tenofovir 245mg) one tablet once daily, or Truvada (tenofovir 245mg/emtricitabine 200mg) or Kivexa (abacavir 600mg/lamivudine 300mg) one tablet once daily plus efavirenz 600mg one tablet once daily for 4 weeks. At week 4, efavirenz is switched to Dolutegravir 50mg (one tablet) once daily
  Interventions: Drug: Dolutegravir, efavirenz, efavirenz/emtricitabine/tenofovir

INTERVENTIONS:
Drug: Dolutegravir, efavirenz, efavirenz/emtricitabine/tenofovir — Arm 1: Switch efavirenz to dolutegravir immediately (at baseline) for 12 weeks Arm 2: Continue on pre-study regimen (unchanged) for 4 weeks and then switch efavirenz to dolutegravir for 12 weeks
  Other Names: Tivicay®, efavirenz, Atripla®

SUMMARY:
This is a phase IV, open label, multicentre trial that will be taking place at 4 sites in the United Kingdom (UK). Efavirenz which is taken in combination with Kivexa® or as part of the combination pill, Atripla® is a recommended firstline regimen for the treatment of Human Immunodeficiency Virus-1 (HIV- 1) infection. Treatment against the HIV virus is also referred to as antiretroviral therapy.

Toxicity is the most common reason for modification of firstline therapy. Central Nervous System (CNS) side effects such as difficulty with sleeping & bad dreams are common side effect of Efavirenz based therapy and is one of the most frequent reasons for switching or discontinuing highly active antiretroviral therapy.

Dolutegravir is within a novel class of antiretroviral agents licensed in the UK for the treatment of HIV. In combination with Truvada®, it showed fewer side effects when compared to Efavirenz in other clinical studies, where patients were starting HIV treatment for the first time, or switching from other agents.

The purpose of the study is to investigate the benefits of switching away from Eefavirenz (in combination with Kivexa® or as part of the combination pill, Atripla®) to Dolutegravir in patients with CNS side effects (such as difficulty with sleeping, bad dreams etc).

DETAILED DESCRIPTION:
The main aim of this study is to investigate the benefits of switching from Efavirenz (taken in combination with Kivexa®or as part of the combination pill, Atripla®) in patients with Central Nervous System (CNS) side effects (such as difficulty with sleeping, bad dreams etc). The study aims to investigate the effect of switching Efavirenz to Dolutegravir while continuing Truvada (tenofovir plus emtricitabine, two constituents of Atripla) or Kivexa. Dolutegravir will be the only new component of the combination.

In addition to the aims stated above, the study also aims:

To investigate whether switching to dolutegravir based combination Antiretroviral Therapy (cART) is associated with resolution of CNS toxicity (determined by CNS questionnaire) at 12 weeks post switch To investigate continued virological suppression at levels of <400 and <50 copies/ml in individuals switching to dolutegravircontaining cART at 4 and 12 weeks post switch To investigate changes in cluster of differentiation 4+ (CD4+) cell count in individuals switching to dolutegravircontaining cART over 12 weeks post switch To investigate the safety (laboratory and non CNS adverse events) of switching to dolutegravir based cART over 12 weeks post switch To investigate changes in quality of life in individuals switching to dolutegravir based cART as assessed by Quality of life (EuroQOL) questionnaires over 12 weeks post switch To investigate the impact of switching to dolutegravir based CART on anxiety and depression (as determined by Hospital Anxiety and Depression Score (HADS) over 12 weeks post switch To investigate changes in quality of sleep in individuals switching to dolutegravir based cART as per standardized sleep questionnaire at 4 and 12 weeks post switch To assess the impact of switching to dolutegravir based cART on adherence by standard questionnaire over 12 weeks post switch To investigate changes in neuropsychiatric function in individuals switching to dolutegravir based cART by CogState battery and Instrumental Activities of Daily Life (IADL) questionnaire over 12 weeks post switch To investigate changes in fasting cholesterol and triglycerides in individuals switching to dolutegravir based cART over 12 weekspost switch To investigate Efavirenz (EFV) plasma decay and its impact on Dolutegravir (DTG) concentrations following the switch (Maximum Concentration (Cmax), Minimum Concentration (Cmin), Area Under the concentration-time Curve (AUC) at weeks 1, 2 and 3 post switch) To investigate the association between genetic polymorphisms in drug disposition genes and drug exposure To assess changes in the levels of tryptophan, kynurenine, kynurenine/tryptophan ratio, neopterin, tumour necrosis factorα and interferonγ in plasma following treatment switch from efavirenz to dolutegravir.

To investigate the relationship between the immune activation biomarkers and the kynurenine/tryptophan ratio at baseline and post switch.

To investigate the relationship between the kynurenine/tryptophan ratio and measures of CNS toxicity and neurocognitive impairment at baseline and postswitch.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female aged 18 years or older
* Has HIV-1 infection documented in their medical notes
* Has signed the Informed Consent Form voluntarily
* Is willing to comply with the protocol requirements
* Is currently on an antiretroviral regimen comprising at least three licensed antiretroviral agents one of which is EFV, for at least 12 weeks
* No previous exposure to integrase inhibitors
* Has an HIV-plasma viral load at screening <400 copies/mL (single re-test allowed)
* Has a CD4 cell count at screening >50 cells/mm3
* Estimated glomerular filtration rate (MDRD) >50 ml/min.
* Has symptomatic CNS related toxicity associated with EFV at least Grade 2 by ACTG criteria
* If female and of childbearing potential, is using effective birth control methods (as agreed by the investigator) and is willing to continue practising these birth control methods during the trial and for at least 30 days after the end of the trial.

Exclusion Criteria:

* Infected with HIV-2
* Using any concomitant therapy disallowed as per SPC for the study drugs
* Has acute viral hepatitis including, but not limited to, A, B, or C
* Subjects positive for Hepatitis B at screening (+HBsAg), or anticipated need for Hepatitis C virus (HCV) therapy during the study
* Alanine aminotransferase (ALT) greater than or equal to 5 times the upper limit of normal (ULN), OR ALT greater than or equal to 3xULN and bilirubin greater than or equal to 1.5xULN (with >35% direct bilirubin)
* Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Any investigational drug within 30 days prior to the trial drug administration
* Has received dolutegravir in the past
* Any clinical evidence of baseline resistance mutations
* History or presence of allergy to DTG or excipients (D-Mannitol, Microcystalline Cellulose, Povidone, Croscarmellose Sodium, Sodium Stearyl Fumarate, Talc, white film coat)
* Subjects with moderate to severe hepatic impairment (Class B or greater) as determined by Child-Pugh classification
* Moderate or severe renal impairment (creatinine clearance < 50ml/min by Cockroft-Gault method)
* If female, she is pregnant or breastfeeding
* Screening blood result with any grade 3/4 toxicity according to Division of AIDS (DAIDS) grading scale, except: asymptomatic grade 3 glucose, amylase or lipid elevation or asymptomatic grade 4 triglyceride elevation (re-test allowed).
* Any condition (including drug/alcohol abuse) or laboratory results which, in the investigator's opinion, interfere with assessments or completion of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-03 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Rate of neuropsychiatric and central nervous system (CNS) toxicity | 4 weeks post switch, day1
  The rate of neuropsychiatric and central nervous system (CNS) toxicity (as measured by a questionnaire based on EFV Summary of Product Characteristics (SPC) and graded based on the ACTG adverse event scale) after 4 weeks of dual N(t)RTI plus DTG therapy:
  * Sum total of all grades of CNS adverse events
  * Median number of AIDS Clinical Trial Group (ACTG) grade 2-3 CNS adverse events Results 4 weeks post switch for each arm will be compared with baseline results and week 4 results will be compared between arms (ie 4 weeks post switch for arm 1 and day of switch for arm 2.).

SECONDARY OUTCOMES:
Rate of neuropsychiatric and central nervous system (CNS) toxicity | 12 weeks post switch, day1
  The rate of neuropsychiatric and central nervous system (CNS) toxicity (as measured by a questionnaire based on EFV SPC and graded based on the ACTG adverse event scale) after 12 weeks of dual Nucleoside/Nucleotide Reverse Transcriptase Inhibitor (N(t)RTI) plus DTG therapy:
  * Proportion of subjects with ACTG grade 2-3 events
  * Sum total of all grades of CNS adverse events
  * Median number of ACTG grade 2-3 CNS adverse events Results 12 weeks post switch for each arm will be compared with baseline results.
Virologic suppression | 4 and 12 weeks post switch, day1
  • Proportion of subjects maintaining virologic suppression to <50 and <400 copies/ml, 4 and 12 weeks post switch to dual N(t)RTI plus DTG
CD4 cell count and % | 4 and 12 weeks post switch, day1
  Change in CD4 cell count and % from baseline compared with 4 and 12 weeks post switch to dual N(t)RTI plus DTG
Quality of life | 4 and 12 weeks post switch, day1
  Changes in quality of life as assessed by Quality of life EuroQOL questionnaires at baseline, 4 and 12 weeks post switch
CNS toxicity | 4 and 12 weeks post switch, day1
  Change from baseline of CNS toxicity as measured by Hospital Anxiety and Depression (HADS) score at 4 and 12 weeks post switch to dual N(t)RTI plus DTG therapy, each compared with baseline
Sleep | 4 and 12 weeks post switch, day1
  Change in sleep from baseline compared with weeks 4 and 12 post switch to dual N(t)RTI plus DTG therapy, as determined by the Pittsburgh Sleep Score
Adherence | 4 and 12 weeks post switch, day1
  Change from baseline in adherence after 4 and 12 weeks of dual N(t)RTI plus DTG therapy as measured by the Medication Adherence Self-Report Inventory (M-MASRI) questionnaire
Neurocognitive assessment | 4 and 12 weeks post switch, day1
  Change from baseline in NeuroCognitive (NC) function after 4, and 12 weeks of dual N(t)RTI plus DTG therapy as determined by computerised NC assessment (CogState) and Instrumental Activities of Daily Life (IADL) questionnaire
Cholestrol levels | 4 and 12 weeks post switch, day1
  Change from baseline in median fasting cholesterol (total, HDL, LDL and total:HDL ratio) and triglycerides after switching to dual N(t)RTI plus DTG therapy at 4 and 12 weeks post switch
Laboratory values | 4 and 12 weeks post switch, day1
  Proportion of patients with grade 2-4 laboratory parameters (excluding lipids) after 4 and 12 weeks of dual N(t)RTI plus DTG therapy compared with baseline and proportion of patients with grade 2-4 non-CNS adverse events after 4 and 12 weeks of dual N(t)RTI plus DTG therapy compared with baseline
Efavirenz plasma concentration and Dolutegravir pharmacokinetics | 1, 2 and 3 weeks post switch, day1
  Efavirenz plasma concentration decay and DTG Pharmacokinetics (PK) (Cmax, Cmin, AUC) at weeks 1, 2 and 3 post switch
Protein levels | 12 weeks post switch, day1
  To assess changes in the levels of Triptophan (TRP), Kynurenic (KYN), KYN/TRP ratio, neomycin (NEO), Tumor Necrosis Factor (TNF-α) and Interferon (IFN-γ) in plasma at baseline/time of switch and 12 wks post-switch for all patients.
Difference in protein levels between the 2 arms | 12 weeks post switch, day1
  To assess differences between the immediate switch and delayed switch groups with regards to changes in the levels of TRP, KYN, KYN/TRP ratio, NEO, TNF-α and IFN-γ in plasma at baseline/time of switch and 12 wks post-switch
Relationship between immune activation markers and protein ratio | Baseline and post switch, day1
  To investigate the relationship between the IA biomarkers and the KYN/TRP ratio at baseline and post-switch.
Relationship between protein ratio and CNS toxicity and neurocognitive impairment | Baseline and post switch, day1
  To investigate the relationship between the KYN/TRP ratio and measures of CNS toxicity and NCI at baseline and post-switch.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Nelson, MD, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- Chelsea and Westminster Hospital, London, United Kingdom